CLINICAL TRIAL: NCT03457415
Title: Collection of Sputum and Sputum Labeling Utilizing Synthetic Meso-Tetra (4-Carboxyphenyl) Porphyrin (TCPP) for Detection of Lung Cancer
Brief Title: Collection of Sputum and Labeling for Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: bioAffinity Technologies Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BA-002
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
Keywords: LDCT; Sputum; High-risk Smoker; Porphyrin; Early detection
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Cohort: Healthy Cohort: current non-smoker who has smoked less than 5 pack-years in his or her lifetime, and if smoked, quit more than 15 years ago, and has no known lung disease.
- High-risk Cohort: High-risk Cohort: individual aged ≥55-74 who is a current smoker with a smoking history of at least 30 pack-years or current non-smoker who has a smoking history of at least 30 pack-years and quit smoking within the past 15 years.
- Cancer Cohort: Cancer Cohort: individual who has been diagnosed by a physician as highly suspect for having lung cancer, but has not yet undergone a biopsy nor received therapy, and after providing a sputum sample is confirmed to have lung cancer by biopsy.

SUMMARY:
The primary objective of this study is to compare Assay results to diagnoses determined by currently accepted standards for lung cancer detection. This will be accomplished by analysis of sputum samples from three cohorts including healthy Participants, high risk Participants, and cancer patient Participants using the Assay as developed in accordance with findings of bioAffinity protocol BA-001 to confirm assay results. Adjustments will be made as necessary to finalize Assay design for clinical trials and commercialization.

The secondary objective of this study is to determine optimum methods for collection of sputum samples. Three sputum collection methods used by high risk Participants will be compared. Individuals at high risk for lung cancer will be assigned to one of three sputum collection cohorts including (1) acapella® airway assist device under medical supervision to obtain a single sputum sample; (2) acapella® airway assist device to obtain a sputum sample over a three-day period, and (3) individuals who under medical supervision will collect a single sputum sample assisted by nebulization of between 0.9% to 10% hypertonic saline. Samples will be compared to determine the optimal collection method for sample analysis by CyPath® Lung.

DETAILED DESCRIPTION:
This study will be performed at multiple study centers to collect sputum samples from three cohorts including (1) healthy Participants, (2) individuals at high risk for lung cancer and (3) individuals who have been diagnosed with lung cancer. Participants in the high risk cohort will undergo low dose computed tomography (LDCT) scans to confirm they do not have lung cancer. LDCT scans will be evaluated by a radiologist at each site. Each subject's sputum specimen will be processed in accordance with individual experimental protocol at the laboratory of bioAffinity Technologies, Inc. (BA) located at the University of Texas at San Antonio 1604 main campus in San Antonio, Texas, or at the Research DX laboratory in Irvine, California.

Once a sample is obtained and delivered to the laboratory, the Assay methodology consists of chemical dissociation of sputum to produce a single cell suspension sample that is labeled with antibodies to identify various types of cell populations in the sample. Thereafter, sputum samples are stained with the cancer detection compound, CyPath® Lung. This compound has a unique fluorescent spectrum that can be analyzed by a flow cytometer. The flow cytometric analysis confirms that the sample is from the deep lung and identifies various cell populations based on characteristics such as cell size, granularity, and antigen expression. Cancer samples can be distinguished from non-cancer samples by the presence of highly fluorescent cells labeled by CyPath®. In this manner, CyPath® can identify lung cancer cells and other distinguishing cells that have been sloughed off in the lungs and coughed up in the sputum sample, including cancer cells.

Researchers who will be blinded as to the Participant's identity will perform the experiments that compare the characteristics of samples collected by the alternate sample collection methods and labeled by CyPath® Lung. In the latter phase of the study, the analytical results of sputum sample analysis requires that the researchers be blinded to the classification of the sputum sample and methods of collection.

Findings from the CyPath® Lung Assay will not be used in the diagnosis of Participants or subsequent treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria to be enrolled in this study:

* Male or female
* 21 years of age or older
* Willing to provide primary care physician contact information to the investigator and agree to have medical information released if indicated
* Meet requirements of one of three cohorts in the study:

Healthy Cohort: Current non-smoker who has smoked less than 5 pack-years in his or her lifetime, and if smoked, quit more than 15 years ago, and has no known lung disease.

High Risk Cohort: Individual aged ≥55-74 who is a current smoker with a smoking history of at least 30 pack-years, or current non-smoker who has a smoking history of at least 30 pack-years, and quit smoking within the past 15 years.

Cancer Cohort: Individual who has been diagnosed by a physician as highly suspect for having lung cancer but has not yet undergone a biopsy nor received therapy, and after providing a sputum sample is confirmed to have lung cancer by biopsy.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from the study:

* Severe obstructive lung disease and unable to cough with sufficient exertion to produce a sputum sample. Participants with lung disease that are able to cough with sufficient exertion to produce a sputum sample are not excluded from the study
* Angina with minimal exertion
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population:
  Male and female Participants, 21 years of age or older, who meet the requirements of one of three cohorts described below:
  * Healthy Cohort
  * High-risk Cohort
  * Cancer Cohort
  Participants who meet any of the following criteria will be excluded from the study:
  * Severe obstructive lung disease and unable to cough with sufficient exertion to produce a sputum sample due to lung disease. Participants with lung disease that are able to cough with sufficient exertion to produce a sputum sample are not excluded from the study.
  * Currently undergoing treatment for cancer. Participants who are on long-term medications used for treatment and/or prevention of cancer, such as Tamoxifen for breast cancer, are not excluded.
  * Angina with minimal exertion
  * Pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identification of Differential Characteristics | 320 days
  The primary outcome measure is to identify differential characteristics (using flow cytometry for high-throughput screening of Assay labeled sputum samples) between samples taken from healthy Participants, Participants at high risk for lung cancer who are free of the disease, and Participants with confirmed lung cancer.

SECONDARY OUTCOMES:
Sputum Collection Methodology | 320 days
  The secondary endpoint is evaluation of the suitability of sputum samples collected by the three different methods.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Atlantic Respiratory Institute, Summit, New Jersey
  - Radiology Associates of Albuquerque, Albuquerque, New Mexico
  - South Texas Veterans Health Care System (STVHCS)/Audie L. Murphy Memorial Veterans Hospital, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bederka LH, Sanchez JR, Rebeles J, Araujo PR, Grayson MH, Lai SC, DePalo LR, Habib SA, Hill DG, Lopez K, Patriquin L, Sussman R, Humphreys J, Reveles XT, Rebel VI. Sputum analysis by flow cytometry; an effective platform to analyze the lung environment. PLoS One. 2022 Aug 17;17(8):e0272069. doi: 10.1371/journal.pone.0272069. eCollection 2022. PMID 35976857
- [Background] Grayson M, Lai SC, Bederka LH, Araujo P, Sanchez J, Reveles XT, Rebel VI, Rebeles J. Quality-Controlled Sputum Analysis by Flow Cytometry. J Vis Exp. 2021 Aug 9;(174). doi: 10.3791/62785. PMID 34424239
- [Background] Lemieux ME, Reveles XT, Rebeles J, Bederka LH, Araujo PR, Sanchez JR, Grayson M, Lai SC, DePalo LR, Habib SA, Hill DG, Lopez K, Patriquin L, Sussman R, Joyce RP, Rebel VI. Detection of early-stage lung cancer in sputum using automated flow cytometry and machine learning. Respir Res. 2023 Jan 21;24(1):23. doi: 10.1186/s12931-023-02327-3. PMID 36681813